CLINICAL TRIAL: NCT02382562
Title: Brief Behavioral Activation Intervention for Depressed Asthma and Urticaria Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Gailen D. Marshall Jr., MD PhD, Gailen D. Marshall, Jr., MD, PhD, University of Mississippi Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0340
Record Dates: First submitted 2015-03-02; First posted 2015-03-06 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Depression; Asthma; Urticaria
Keywords: Depression; Asthma; Urticaria
MeSH Terms: conditions — Depression; Asthma; Urticaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brief Behavioral Activation Intervention (Experimental): All eligible participants will undergo the Brief Behavioral Activation Intervention.
  Interventions: Behavioral: Brief Behavioral Activation Intervention

INTERVENTIONS:
Behavioral: Brief Behavioral Activation Intervention — Clinical psychologists (investigators) will instruct the participant in ways to become more active in life, particularly with regards to activities that the participant finds pleasurable and meaningful. The intervention will take one hour to complete. Following the intervention, the participant will receive brief, weekly text or email reminders for the next 4 weeks (total of 4) to engage in pleasurable and meaningful activities during the week.

SUMMARY:
Depression and other unhealthy behaviors, such as not taking medication as prescribed and not attending doctor visits have been suggested to increase the worsening of allergic diseases (e.g. asthma, urticaria). We intend to determine whether a one-session behavioral intervention is effective in helping with depression and controlling disease symptoms. We will measure this using pre- and post-intervention surveys.

DETAILED DESCRIPTION:
The purpose of this research study is to investigate whether a one-session behavioral activation intervention for depression can successfully reduce depression and improve asthma or urticaria disease-relevant outcomes (medication adherence, doctor's visits, substance abuse) in clinical patients with asthma or urticaria who report heightened levels of depression and are seen in the UMMC Allergy Clinic.

ELIGIBILITY:
Inclusion Criteria:

* Potential participants should be between the ages 18 and 64, seen in the UMMC Allergy Clinic with either asthma or urticaria and who report symptoms of depression in the previous 2 weeks.

Exclusion Criteria:

* Potential participants younger than 18 and older than 64 or who do not speak English or cannot comprehend the consent form or women who are pregnant are excluded.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2016-10-17 (Actual)

PRIMARY OUTCOMES:
Asthma Control Test | 4 weeks
  Changes in asthma control over a 4 week period.
Urticaria Control Test | 4 weeks
  Changes in urticaria control over a 4 week period.

SECONDARY OUTCOMES:
Asthma Quality of Life Questionnaire | 4 weeks
  Changes in asthma quality of life over a 4 week period.
Urticaria Activity Score Questionnaire | 4 weeks
  Changes in the activity of urticaria over a 4 week period.
Psychological Measures (Composite) | 4 weeks
  Effects of brief behavioral activation intervention based upon psychological differences including depression and anxiety measured over a 4 week period.

OTHER OUTCOMES:
Immune biomarkers | 4 weeks
  Changes in Regulatory T (Treg), Type 1 Regulatory (Tr1), T helper (TH3), T helper 1 (TH1), T helper 2 (TH2), cells, Interferon gamma (IFNg), Interleukin 4 (IL4) and Interleukin 10 (IL10) cytokine production from baseline to 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Gailen D Marshall, Jr., MD, PhD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center - Allergy, Immunology and Asthma Care Clinic, Jackson, Mississippi, United States